CLINICAL TRIAL: NCT01669551
Title: A Phase 1 Feasbility Study Of Volume Intracardiac Echo In Assessment Of Patients With Structural And Valvular Heart Disease Undergoing Percutaneous Transcatheter Therapy
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: UPenn 815656
Record Dates: First submitted 2012-08-16; First posted 2012-08-21 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2012-08

CONDITIONS: Structural and Valvular Heart Disease
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Structural or Valvular Heart Disease

SUMMARY:
This study will compare 3 dimensional intracardiac echo (ICE) with 2 dimensional ICE or transesophageal echo in patients with structural and valvular heart disease who are already scheduled to undergo a percutaneous intervention. Specifically those patients would be those scheduled for a PFO or ASD repair, mitral balloon valvuloplasty, diagnostic cardiac catheterization assessment of aortic stenosis and those undergoing transcatheter aortic valve replacement.

ELIGIBILITY:
Inclusion Criteria:

* patients in the study population referred to the cardiac catheterization laboratory for a percutaneous procedure to treat structural or valvular heart disease

Exclusion Criteria:

* Class IV CHF, inadequate femoral access, coagulation abnormalities, intracariac thrombus or DVT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with structural or valvular heart disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Comparison of volume intracardiac echo imaging to 2 dimensional echo | Comparison study

CONTACTS AND LOCATIONS:
Overall Officials: Howard Herrmann, M.D., Principal Investigator — University of Pennsylvania

REFERENCES:
- [Derived] Silvestry FE, Kadakia MB, Willhide J, Herrmann HC. Initial experience with a novel real-time three-dimensional intracardiac ultrasound system to guide percutaneous cardiac structural interventions: a phase 1 feasibility study of volume intracardiac echocardiography in the assessment of patients with structural heart disease undergoing percutaneous transcatheter therapy. J Am Soc Echocardiogr. 2014 Sep;27(9):978-83. doi: 10.1016/j.echo.2014.04.022. Epub 2014 Jun 11. PMID 24930123
- [Derived] Kadakia MB, Silvestry FE, Herrmann HC. Intracardiac echocardiography-guided transcatheter aortic valve replacement. Catheter Cardiovasc Interv. 2015 Feb 15;85(3):497-501. doi: 10.1002/ccd.25409. Epub 2014 Feb 10. PMID 24478152